CLINICAL TRIAL: NCT04463082
Title: Assessment of the Current State of Volume Status in Children by Ultrasound Measurement of Vena Cava Inferior and Vena Jugularis Interna Combined With Passive Leg Raise: a Pilot Study
Brief Title: Non-invasive Assessment of the Current State of Hydration in Children by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-OPRIP-US-fluids
Record Dates: First submitted 2020-06-15; First posted 2020-07-09 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Gastroenteritis; Diabetes Mellitus (Ketoacidosis)
Keywords: children; dehydration; ultrasound; vena cava inferior; vena jugularis; passive leg raise
MeSH Terms: conditions — Gastroenteritis; Diabetes Mellitus; Ketosis; Dehydration

STUDY DESIGN:
Intervention Model Description: The pediatric patients will be divided into three groups, according to weight: 10-20kg, 20-30kg, 30-50kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight category 10-20kg (Experimental): Pediatric patients with a weight of 10-20kg will be enrolled in this arm.
  Interventions: Procedure: Intravenous administration of fluids
- Weight category 20-30kg (Experimental): Pediatric patients with a weight of 20-30kg will be enrolled in this arm.
  Interventions: Procedure: Intravenous administration of fluids
- Weight category 30-50kg (Experimental): Pediatric patients with a weight of 30-50kg will be enrolled in this arm.
  Interventions: Procedure: Intravenous administration of fluids

INTERVENTIONS:
Procedure: Intravenous administration of fluids — Intravenous administration of fluids (20ml/kg, but the maximum volume will be limited up to 500ml) within 60 minutes.

SUMMARY:
Children with clinical signs of severe dehydration will be examined by ultrasound in a supine position during admission. Children aged between 1 and 15years will be divided into three weight groups: 10-20kg, 20-30kg, 30-50kg. Early after admission 1st measurement of diameters of vena cava inferior (VCImax, VCImin) during breathing cycles and diameters of both venae jugulares (VJI dx max, min, VJI sin max, min) before and after passive leg raise maneuver will be recorded. After a defined fluid infusion within 60 minutes, a second examination will be evaluated and compared with the first one. The investigators considered also echocardiography to measure CO changes however they wanted to make it as simple as it might be at emergency during the night shift without an experienced cardiologist.

DETAILED DESCRIPTION:
Only children admitted to the hospital with clinically detectable dehydration (weight loss, dry skin, sunken eyes, no tears) will be evaluated. Weight, noninvasive blood pressure measurement, pulse rate will be recorded. Measurements would be performed with an ultrasound probe with a low frequency (2-5 MHz), a curved array transducer will be used. In the supine position, the ultrasound probe will be placed in the substernal area, in the longitudinal and transversal plane, 1 cm caudal to the confluence of the hepatic veins, and it will be operated in M-mode. The largest (VCImax) and smallest (VCImin) diameters will be measured and the collapsibility index will be calculated (according to the formula: VCImax - VCI min / VCI max x100). Immediately after this examination measurement of the right VJImax, min and the left VJImax, min will be measured again in the supine position, then after passive leg raise (lifting the lower limbs 45st. for at least 1minute ) VJImax, min. and left VJImax, min will be measured. The collapsibility index for right and left VJI would be calculated according to the formula: VJImax - VJI min / VJI max x100. After a defined fluid infusion (20ml/kg, but the maximum volume will be limited to 500ml, this means that over 25kg weight we would apply not more than 500ml) within 60 minutes. A control examination of VCI, right VJI, and left VJI will be evaluated the same way as first and compared with the previous one.

ELIGIBILITY:
Inclusion Criteria:

* previously healthy children
* history and clinical signs of dehydration (gastroenteritis, diabetic ketoacidosis)

Exclusion Criteria:

* congenital heart diseases
* intestinal obstruction
* any signs of abdominal hypertension
* any illnesses known to affect the volume status

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in vena cava inferior diameter pre- and post-hydration | 60 minutes
  Change in vena cava inferior diameter (in millimetres) will be measured before and after hydration.
Change in vena jugularis interna diameter pre- and post-hydration (on the right side) | 60 minutes
  Change in vena jugularis interna diameter (in millimetres) will be measured before and after hydration (on the right side).
Change in vena jugularis interna diameter pre- and post-hydration (on the left side) | 60 minutes
  Change in vena jugularis interna diameter (in millimetres) will be measured before and after hydration (on the left side).
Change in collapsibility index pre- and post-hydration | 60 minutes
  Change in collapsibility index values (in per cent) will be measured before and after hydration.

SECONDARY OUTCOMES:
Correlation to body surface area | 60 minutes
  All obtained parameters from the other Outcome Measures will be correlated to the body surface area of the patient (measured in m2)

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Zaoral, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators have no plan to share individual participant data with other researchers; the data will be provided upon a written request.

REFERENCES:
- [Background] Unluer EE, Kara PH. Ultrasonography of jugular vein as a marker of hypovolemia in healthy volunteers. Am J Emerg Med. 2013 Jan;31(1):173-7. doi: 10.1016/j.ajem.2012.07.003. Epub 2012 Sep 11. PMID 22980368
- [Background] Bauman Z, Coba V, Gassner M, Amponsah D, Gallien J, Blyden D, Killu K. Inferior vena cava collapsibility loses correlation with internal jugular vein collapsibility during increased thoracic or intra-abdominal pressure. J Ultrasound. 2015 Sep 18;18(4):343-8. doi: 10.1007/s40477-015-0181-2. eCollection 2015 Dec. PMID 26550073
- [Background] Lu GP, Yan G, Chen Y, Lu ZJ, Zhang LE, Kissoon N. The passive leg raise test to predict fluid responsiveness in children--preliminary observations. Indian J Pediatr. 2015 Jan;82(1):5-12. doi: 10.1007/s12098-013-1303-5. Epub 2013 Dec 11. PMID 24327086